CLINICAL TRIAL: NCT06597331
Title: Prospective Observational Study of Myocardial Stunning in Patients Hospitalized for Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Cardiac Assessment and Takotsubo-stunning Among COPD-exacerbations In-Hospital
Acronym: CATCH
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Rickard Zeijlon, MD, PhD, specialist of internal medicine, Sahlgrenska University Hospital
Other Study IDs: Dnr 2024-02071-01
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Takotsubo Cardiomyopathy; Acute Heart Failure
Keywords: Takotsubo syndrome; COPD; Echocardiography; Screening; Trigger
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, biobanking for later analysis of metabolomics, proteomics, miRNA and mRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective observational study is to investigate to what extent acute exacerbation of chronic obstructive pulmonary disease (AE-COPD) triggers Takotsubo-stunning, and how this affects the outcome for these patients.

The main questions it aims to answer are:

1. What is cumulative incidence of Takotsubo-stunning in patients hospitalized for AE-COPD at Sahlgrenska University Hospital/S (Gothenburg, Sweden)?
2. Among patients hospitalized for AE-COPD at Sahlgrenska University Hospital/S, what is the risk of in-hospital clinical manifestations of acute heart failure in patients with Takotsubo-stunning compared to those without?

DETAILED DESCRIPTION:
PURPOSE

The purpose of Cardiac Assessment and Takotsubo-stunning among COPD-exacerbations in-Hospital (CATCH) is to investigate to what extent AE-COPD triggers Takotsubo-stunning in patients admitted to in-hospital care, and how this affects the outcome for these patients.

BACKGROUND

Acute exacerbation of chronic obstructive pulmonary disease (AE-COPD) may cause acute heart failure due to stress-induced myocardial stunning, which is probably underdiagnosed or undiagnosed in clinical routine. Elements of myocardial stunning is associated with several conditions, however, the Takotsubo syndrome (TS) is probably a pure form of myocardial stunning. Therefore, the term "Takotsubo-stunning" is sometimes used to describe the myocardial stunning that occur in TS.

TS is an acute heart failure syndrome associated with emotional or physical stress predominately affecting females (>90% females) in the postmenopausal ages. TS is characterized by rapid onset of regional wall motion abnormality (typically widespread apical akinesia) and reversible left ventricular dysfunction. One of the most widely reported physical triggers of TS is AE-COPD and COPD is overrepresented among patients with TS. Concurrent respiratory disease such as AE-COPD complicate the diagnosis of TS, since the cardiac condition may be masked by pulmonary symptoms, and the respiratory symptoms may be further exacerbated by Takotsubo-stunning. Also, a cornerstone in the treatment for AE-COPD is high doses of beta-2-adrenergic agonists through inhalation. This may be unfavourable (and possibly detrimental) for a patient with Takotsubo-stunning, since adrenergic overstimulation in general, and overstimulation of cardiac beta-2-adrenergic receptor in particular, seems to be involved in the pathophysiology of TS.

Although it is known that AE-COPD is common among patients with TS, research is lacking regarding the inverse relationship, i.e. how common TS is among patients with AE-COPD. Therefore, the investigators aim to elucidate to what extent AE-COPD triggers Takotsubo-stunning, through investigating the incidence of Takotsubo-stunning in AE-COPD.

HYPOTHESES

1. Among adult patients admitted for in-hospital care for AE-COPD at Sahlgrenska University Hospital/S (Gothenburg, Sweden) a non-negligible proportion (more than one out of ten) develop Takotsubo-stunning as complication triggered by the AE-COPD.
2. Within in the above-mentioned patient group, AE-COPD complicated by Takotsubo-stunning is associated with more clinical signs of acute heart failure and a worse outcome (longer length of stay, more complications, higher mortality) compared to AE-COPD not complicated by TS.

STUDY DESIGN

CATCH is a prospective observational cohort study, originating from the section for Acute and Cardiovascular Medicine at the department of Emergency Medicine and Geriatrics at Sahlgrenska University Hospital/S (SU/S). Patients admitted to SU/S hospital wards 90 or 91 (acute internal medicine); 19 or 32 (pulmonary medicine and general internal medicine); 16 or 29 (endocrinology and gastroenterology) for AE-COPD are eligible for inclusion.

To identify possible Takotsubo-stunning, included patients will be screened for echocardiographic signs of regional wall motion abnormality and/or left ventricular dysfunction, where positive and negative screening will be defined as follows:

POSITIVE: Presence of any regional wall motion abnormality and/or left ventricular dysfunction (LVEF <50%)

NEGATIVE: Absence of regional wall motion abnormality and no left ventricular dysfunction (LVEF >50%)

If negative, screening will be repeated once, after 24 (+/-6) hours. If positive (i.e. screening reveals signs of regional wall motion abnormality and/or cardiac dysfunction), screening will be converted to a full echocardiographic examination according to standard clinical protocol, which will be repeated after 24 (+/-6) hours and after 30 (+/-48 hours) days. Reversibility will be defined as improvement in cardiac function between first positive echocardiographic examination and day 30. Such transient cardiac dysfunction will be regarded as Takotsubo-stunning (provided no other cause has been identified, as per diagnostic criteria for TS). Persistent cardiac dysfunction is a pre-defined exclusion-criteria and therefore these patients will be excluded from the analysis. Patients who turn out positive in screening will be offered inclusion in STAMI-study (Stunning in Takotsubo versus Acute Myocardial Infarction, clinical trials identifier NCT04448639, ongoing since 2020).

OTHER PROCEDURES AND COLLECTION OF DATA

All patients will be interviewed according to a questionnaire regarding presenting symptoms. Blood sampling for analysis of NTproBNP, ECG and chest x-ray will be performed at inclusion (day 0) and day 1. Baseline characteristics will be collected from the patients' medical charts and vital parameters will be registered the first three days. In-hospital complications/death will be registered consecutively. COPD GOLD (Global initiative for Obstructive Lung Disease) grade/group and severity of exacerbation will be registered. In follow-up, data from re-evaluation of COPD (clinical routine after hospital care for AE-COPD) will be collected (Spirometry, diffusion capacity, static lung volumes, 6-min walk test. COPD assessment test).

PRIMARY ENDPOINTS

1. 1-year cumulative incidence of Takotsubo-stunning
2. Clinical signs of acute heart failure during hospitalization (defined as modified Killip Class >1, explained below)

Modified Killip Class: To assess clinical signs heart failure, the investigators will use a modified version of Killip Classification of acute heart failure (originally developed for assessing acute heart failure after myocardial infarction). Killip class I-III will be assessed using pulmonary ultrasound instead of auscultation sounds, Killip Class IV (cardiogenic shock) will be assessed unmodified according to clinical routine.

SECONDARY ENDPOINTS

1. In-hospital Major Adverse Cardiac Events (MACE): nonfatal myocardial infarction, nonfatal stroke or cardiovascular death
2. Admission to intensive care unit
3. In-hospital death and death within one year

SCIENTIFIC IMPORTANCE

A link seems to exist between AE-COPD and myocardial stunning/TS. This is important for two main reasons:

1. The cardiac condition may be masked by the respiratory symptoms and the clinical signs of AE-COPD, leading to delayed or missed diagnosis of the cardiac component
2. Myocardial stunning with cardiac dysfunction may further exacerbate the patient's condition, leading to prolonged time to recovery due to concomitant untreated AHF; and an increased risk of severe cardiac complications

Another important aspect is the treatment for AE-COPD, which may include treatment with high doses of beta-2-agonists. Catecholamines are part of the pathophysiological cause of myocardial stunning, and catecholaminergic drugs may further aggravate myocardial stunning. In fact, beta-2-agonists specifically has been shown to likely trigger myocardial stunning/TS. Therefore, the routine treatment for AE-COPD may be associated with a risk of harming patients with concomitant AE-COPD and myocardial stunning. If successful, the CATCH-study may improve the quality of care and outcome for patients with AE-COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) admitted to hospital ward for AE-COPD
* Inclusion within 72 hours of admission,
* Written informed consent

Exclusion Criteria:

* Prior acute myocardial infarction or known pre-existing persistent regional wall motion abnormality or left ventricular dysfunction (left ventricular ejection fraction [LVEF] <50%)
* Expected inability to comply with the protocol (e.g. dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to hospital ward for AE-COPD within 72 hours
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Reversible left ventricular dysfunction (myocardial stunning) according to echocardiography | 30 days
  Echocardiographic signs of myocardial stunning/Takotsubo-stunning at inclusion (day 0) with recovery of left ventricular function at day 1 and/or day 30
Clinical signs of acute heart failure at inclusion (day 0) or day 1 according to the Killip Classification | 2 days
  Acute heart failure will be defined as modified Killip Class >1, and will be compared between patients with vs without myocardial stunning/Takotsubo-stunning

SECONDARY OUTCOMES:
In-hospital Major Adverse Cardiac Events (MACE) | At discharge from hospital (on average 5 days)
  Defined as nonfatal myocardial infarction, nonfatal stroke or cardiovascular death; at some point during hospitalization. Comparison between patients with versus without myocardial stunning/Takotsubo-stunning.
Admission to intensive care unit (ICU) during index hospitalization | At discharge from hospital (on average 5 days)
  Admission to ICU at any point during hospitalization. Comparison between patients with versus without myocardial stunning/Takotsubo-stunning.
In-hospital death and death within one year | At time of in-hospital death or at discharge from hospital (on average 5 days) and after 1 year
  In-hospital death and death within one year. Comparison between patients with versus without myocardial stunning/Takotsubo-stunning.

CONTACTS AND LOCATIONS:
Overall Officials: Rickard Zeijlon, M.D. PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Emergency Medicine and Geriatrics, Sahlgrenska University Hospital/S, Gothenburg, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No